CLINICAL TRIAL: NCT02896582
Title: Phase II Study to Evaluate the Efficacy of Upfront Obinutuzumab in Mantle Cell Lymphoma Patients Treated by DHAP Followed by Autologous Transplantation Plus Obinutuzumab Maintenance Then MRD Driven Maintenance
Brief Title: Efficacy of Upfront and Maintenance Obinutuzumab in Mantle Cell Lymphoma Treated by DHAP and MRD Driven Maintenance
Acronym: LyMa101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LyMa101
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obinutuzumab; Dexamethasone; Cytarabine; Cisplatin; Etoposide; Melphalan; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction - ASCT - maintenance (Experimental): Induction : 4 cycles of GA-DHAP every 21 days - Conditioning regimen and ASCT: GA-BEAM + Autologous transplantation - Maintenance : Obinutuzumab every 2 months for 3 years then every month for patients with positive MRD
  Interventions: Drug: Obinutuzumab; Drug: Dexamethasone; Drug: Aracytine; Drug: Cisplatinum; Drug: Etoposide; Drug: Melphalan; Drug: Carmustine

INTERVENTIONS:
Drug: Obinutuzumab — 1000 mg D1, D8, D15 in GA-DHAP 1000 mg D-8 in GA-BEAM 1000 mg every 2 months for 3 years then every month if MRD+
  Other Names: GA; GA101
Drug: Dexamethasone — 40 mg D1 to D4 in GA-DHAP
Drug: Aracytine — 2g/m² D1 & D2 in GA-DHAP 400 mg/m² D-6 to -3 in GA-BEAM
  Other Names: Cytarabine
Drug: Cisplatinum — 100 mg/m² D1 in GA-DHAP
Drug: Etoposide — 400 mg/m² D-6 to D-3 in GA-BEAM
Drug: Melphalan — 140 mg/m² D-2 in GA-BEAM
Drug: Carmustine — 300 mg/m² D-7 in GA-BEAM
  Other Names: BiCNU; BCNU

SUMMARY:
This study is a multicentric, single arm phase II trial to evaluate the efficacy of upfront obinutuzumab in mantle cell lymphoma patients treated by Cisplatinum-Cytarabine-Dexamethasone (DHAP) followed by autologous transplantation plus obinutuzumab maintenance then Molecular Residual Disease (MRD) driven maintenance

DETAILED DESCRIPTION:
Patients will be recruited over 2 years. They must have a histologically proven diagnosis of mantle cell lymphoma, be aged from 18 to 65 years at the time of registration. Patients must be eligible for autologous transplant and not previously treated for their lymphoma at inclusion. Patients will receive 4 cycles of Obinutuzumab (GA101) and Cisplatinum-Cytarabine-Dexamethasone (GA-DHAP) every 21 days followed by Autologous Stem Cell Transplant (ASCT) using a GA101-Carmustine- Etoposide- Cytarabine- Melphalan (GA-BEAM) conditioning regimen plus a Obinutuzumab maintenance for 3 years then a Obinutuzumab maintenance on demand according to MRD status. Stem cells will be collected after cycle 3 and/or 4 of GA-DHAP.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and age ≤ 65
* Histologically confirmed (according to the World Health Organization (WHO) classification) mantle cell lymphoma. The diagnosis has to be confirmed by phenotypic expression of CD5, CD20 and cyclin D1 or the t(11;14) translocation.
* Bone marrow aspiration performed at inclusion for MRD analyses
* Eligible for autologous stem cell transplant
* Previously untreated MCL
* Stage Ann Arbor II-IV in need of treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Life expectancy of more than 3 months
* Written informed consent
* Patient affiliated by any social security system

Exclusion Criteria:

* Severe cardiac disease: York Heart Association (NYHA) grade 3-4
* Impaired liver (ALanine Amino Transferase (ALAT)/ASparagin Amino Transferase (ASAT) ≥ 2.5 Upper Limit of Normal (ULN), bilirubin ≥ 1.5 ULN), renal (calculated creatinine clearance < 50 ml/min) or other organ function which will interfere with the treatment, if not related to lymphoma.
* History of chronic liver disease
* Hepatic veno-occlusive disease or sinusoidal obstruction syndrome
* Any of the following laboratory abnormalities, if not result of a BM infiltration:
* Absolute Neutrophils Count (ANC) <1,500 /mm3 (1.5 x 109/L)
* Platelet counts < 75,000/mm3 (75 x 109/L)
* Pregnancy/Nursing mothers
* Fertile men or women of childbearing potential unless:
* surgically sterile or ≥ 2 years after the onset of menopause
* willing to use a highly effective contraceptive method
* Patients with a malignancy that has been treated but not with curative intent, unless the malignancy has been in remission without treatment for ≥ 5 years prior to enrollment. Patients with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix are eligible.
* Known seropositivity for Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or other active infection uncontrolled by treatment.
* Viral infection with hepatitis B virus (HBV) defined as hepatitis B surface antigen (HBsAg) positive and/or Hepatitis B core antibody (anti-HBc) positive Note: Patients who are immune due to hepatitis B vaccination or natural infection (HBs Ag and anti-HBc negative, anti-HBs positive) are eligible. But the patients who are immune due to hepatitis B natural infection should consult liver disease experts before start of treatment and should be monitored and managed following local medical standards to prevent hepatitis reactivation
* Prior history of Progressive Multifocal Leukoencephalopathy (PML)
* Vaccination with a live vaccine a minimum of 28 days prior to inclusion (Prolonged B cell depletion)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies. Known sensitivity or allergy to murine products
* Psychiatric illness or condition which could interfere with their ability to understand the requirements of the study.
* Person deprived of his/her liberty by a judicial or administrative decision
* Person hospitalized without consent
* Adult person under legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Molecular Residual Disease (MRD) in bone marrow after 4 cycles of GA-DHAP | 4 cycles (1 cycle is 21 days)
  to evaluate the efficacy of upfront Obinutuzumab (GA101) at the molecular level (MRD) in bone marrow after induction in patients with previously untreated Mantle Cell Lymphoma (MCL) treated by DHAP

SECONDARY OUTCOMES:
Response according to Cheson 99 | 5.5 years (2.5 years of treatment and 3 years of maintenance)
  Response after 2.5 years of treatment and 3 years of maintenance will be evaluated. Assessment of response will be based on the International Workshop to Standardize Response criteria for Non Hodgkin Lymphoma (NHL) (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 1999)
Overall response rate (ORR) | 5.5 years (2.5 years of treatment and 3 years of maintenance)
  Response after 2.5 years of treatment and 3 years of maintenance will be evaluated. Assessment of response will be based on the International Workshop to Standardize Response criteria for NHL (Criteria for evaluation of response in Non-Hodgkin's lymphoma (Cheson, 1999)
Positron Emission Tomography (PET) result | 5.5 years (2.5 years of treatment and 3 years of maintenance)
  PET result after 2.5 years of treatment and 3 years of maintenance will be evaluated. Assessment of PET will be based on Lugano 2014 criteria (according to Cheson & al. Journal of Clinical Oncology 2015).
MRD | 5.5 years (2.5 years of treatment and 3 years of maintenance)
  Molecular residual disease (MRD) after 2.5 years of treatment and 3 years of maintenance will be evaluated. Assessment of MRD will be based on molecular level in bone marrow (BM) according to the European Mantle Cell Lymphoma network (EU-MCL) guidelines.
MRD and after maintenance "on demand" | 8.5 years (2.5 years of treatment and 2x3 years of maintenance)
  Molecular residual disease (MRD) after maintenance "on demand" will be evaluated. Assessment of MRD will be based on molecular level in BM according to EU MCL network guidelines.
Progression Free Survival (PFS) | 8.5 years (2.5 years of treatment and 2x3 years of maintenance)
  PFS is defined as the time from inclusion into the study to the first observation of documented disease progression or death due to any cause. If a subject has not progressed or died, PFS will be censored at the time of last visit with adequate assessment.
Overall survival (OS) | 8.5 years (2.5 years of treatment and 2x3 years of maintenance)
  OS will be measured from the date of inclusion to the date of death from any cause. Alive patients will be censored at their last contact date
Number of patients for whom stemm cell collection will fail | 3 years
  Stem cell collection failure will be evaluated after induction treatment
Duration of MRD negativity | 8.5 years (2.5 years of treatment and 2x3 years of maintenance)
  Duration of MRD negativity is defined as the time from the date of attainment the first negative MRD to the date of positive MRD. Duration or MRD negativity would be assessed for patients with at least one MRD negativity and as survival endpoint.
Treatment duration | 9 years
Average dose | 9 years
Number of premature treatment discontinuation | 9 years
Frequency of premature treatment discontinuation | 9 years
Number of study discontinuation | 9 years
Frequency of study discontinuation | 9 years
Number of adverse events | 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Le Gouill, Pr, Principal Investigator — Nantes University Hospital; Olivier Hermine, Pr, Principal Investigator — Hopital Necker - Paris
Locations (30):
- France (30):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CH d'Avignon, Avignon
  - CHU de Caen, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - CHU de Grenoble, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - CHU Limoges, Limoges
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hôpital Saint Louis, Paris
  - APHP - Hopital Necker, Paris
  - CH Perpignan, Perpignan
  - CHU de Haut Leveque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier Annecy-Genevois, Pringy
  - CHU Robert Debré, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie de Loire, Saint-Priest-en-Jarez
  - CHU de Strasbourg, Strasbourg
  - I.U.C.T Oncopole, Toulouse
  - CHRU Bretonneau, Tours
  - CHU de Brabois, Vandœuvre-lès-Nancy
  - Gustave Roussy Cancer Campus, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarkozy C, Callanan M, Thieblemont C, Oberic L, Burroni B, Bouabdallah K, Damaj G, Tessoulin B, Ribrag V, Houot R, Morschhauser F, Griolet S, Joubert C, Cacheux V, Delwail V, Safar V, Gressin R, Cheminant M, Delfau-Larue MH, Hermine O, Macintyre E, Le Gouill S. Obinutuzumab vs rituximab for transplant-eligible patients with mantle cell lymphoma. Blood. 2024 Jul 18;144(3):262-271. doi: 10.1182/blood.2024023944. PMID 38669626
- [Derived] Bodet-Milin C, Morvant C, Carlier T, Frecon G, Tournilhac O, Safar V, Kraeber-Bodere F, Le Gouill S, Macintyre E, Bailly C. Performance of baseline FDG-PET/CT radiomics for prediction of bone marrow minimal residual disease status in the LyMa-101 trial. Sci Rep. 2023 Oct 24;13(1):18177. doi: 10.1038/s41598-023-45215-y. PMID 37875524
- [Derived] Le Gouill S, Beldi-Ferchiou A, Alcantara M, Cacheux V, Safar V, Burroni B, Guidez S, Gastinne T, Canioni D, Thieblemont C, Maisonneuve H, Bodet-Milin C, Houot R, Oberic L, Bouabdallah K, Bescond C, Damaj G, Jaccard A, Daguindau N, Moreau A, Tilly H, Ribrag V, Delfau-Larue MH, Hermine O, Macintyre E. Molecular response after obinutuzumab plus high-dose cytarabine induction for transplant-eligible patients with untreated mantle cell lymphoma (LyMa-101): a phase 2 trial of the LYSA group. Lancet Haematol. 2020 Nov;7(11):e798-e807. doi: 10.1016/S2352-3026(20)30291-X. Epub 2020 Sep 21. PMID 32971036
- [Derived] Bailly C, Carlier T, Berriolo-Riedinger A, Casasnovas O, Gyan E, Meignan M, Moreau A, Burroni B, Djaileb L, Gressin R, Devillers A, Lamy T, Thieblemont C, Hermine O, Kraeber-Bodere F, Le Gouill S, Bodet-Milin C. Prognostic value of FDG-PET in patients with mantle cell lymphoma: results from the LyMa-PET Project. Haematologica. 2020 Jan;105(1):e33-e36. doi: 10.3324/haematol.2019.223016. Epub 2019 Aug 1. No abstract available. PMID 31371411

DOCUMENTS (2):
  • Study Protocol (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT02896582/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-09): https://cdn.clinicaltrials.gov/large-docs/82/NCT02896582/SAP_001.pdf